CLINICAL TRIAL: NCT00016224
Title: Phase II Trial of Thalidomide in Patients With Ovarian Cancer
Brief Title: Thalidomide in Treating Patients With Refractory or Resistant Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 01-006; CDR0000068611 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-1943
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Thalidomide

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
RATIONALE: Drugs such as thalidomide may stop the growth of cancer cells by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of thalidomide in treating women who have epithelial ovarian cancer that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the time to progression of disease in patients with platinum-refractory or resistant ovarian epithelial carcinoma treated with thalidomide.
* Evaluate the quality of life of patients treated with this regimen.

OUTLINE: Patients receive oral thalidomide once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then every 4 weeks.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study within 9-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial carcinoma
* Platinum-refractory or resistant disease

  * At least 1 prior non-platinum chemotherapy agent required
* Prior bilateral salpingo-oophorectomy and hysterectomy required
* Bidimensionally measurable disease OR CA-125 greater than 100 units/mm3

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Karnofsky 70-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin normal
* AST no greater than 2.5 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 50 mL/min

Other:

* No other prior malignancy except non-melanoma skin cancer unless curatively treated with no evidence of disease within the past 5 years and at low risk for recurrence
* No other clinical circumstances that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy and recovered
* No prior thalidomide

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior cytotoxic therapy and recovered

Endocrine therapy:

* At least 4 weeks since prior hormonal therapy and recovered

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior major surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spriggs, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States